CLINICAL TRIAL: NCT04740619
Title: Natural Orifice Specimen Extraction in Sigmoid Volvulus Patients
Brief Title: Natural Orifice Specimen Extraction in Sigmoid Volvulus
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Ufuk Uylas, Primary investigator, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 2020/178
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Mortality; Morbidity
Keywords: colon; volvulus; natural orifice; laparoscopy; sigmoid
MeSH Terms: conditions — Intestinal Volvulus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Natural Orifice Specimen Extraction — Natural Orifice Specimen Extraction via transanal

SUMMARY:
Sigmoid resection can be performed using conventional and laparoscopic methods. There are few publications in the literature reporting specimen removal from the natural hole in patients with a diagnosis of sigmoid volvulus. Here, the investigators aimed to present the literature that transanal specimen removal is a technically feasible method after laparoscopic surgery in patients with sigmoid volvulus.

DETAILED DESCRIPTION:
Sigmoid resection can be performed using conventional and laparoscopic methods. There are few publications in the literature reporting specimen removal from the natural hole in patients with a diagnosis of sigmoid volvulus. Here, the investigators aimed to present the literature that transanal specimen removal is a technically feasible method after laparoscopic surgery in patients with sigmoid volvulus. The documents of patients who were operated on for sigmoid volvulus between 2018 and 2019 were retrospectively reviewed. Patients who had been used transanal for specimen extraction by elective laparoscopic sigmoid colon resection were included in the study. Patients' gender, age, comorbidity, operation time, operative difficulties, complications, length of stay, and mortality findings were analyzed. Laparoscopic sigmoid resection and transanal specimen removal were performed in eight patients. Specimen extraction surgery from the natural hole is increasingly preferred. the investigators think that natural hole surgery can be performed more easily and reliably in sigmoid volvulus due to the large diameter of the colon.

ELIGIBILITY:
Inclusion Criteria:

* transanal for specimen extraction by elective laparoscopic sigmoid colon resection

Exclusion Criteria:

* emergency surgery
* conventional open sigmoid resection
* conventional laparoscopic sigmoid resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sigmoid volvulus patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
mortality | 1 year
  mortality after this procedure
morbidity | through study completion, an average of 1 year
  morbidity after this procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No